CLINICAL TRIAL: NCT04957563
Title: Clinical Utility of Olfactory Rehabilitation: Treatment for Pacients With Neurosensorial Anosmia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cristina Gomez Calero (Other)
Responsible Party: Sponsor-Investigator, Cristina Gomez Calero, PhD. Professor. Occupational therapist, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09/79 (HUFA)
Record Dates: First submitted 2021-06-09; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Anosmia; Occupational Therapy; Brain Injuries, Traumatic
Keywords: occupational therapy; anosmia; brain injuries, traumatic
MeSH Terms: conditions — Anosmia; Brain Injuries, Traumatic | interventions — Olfactory Training

STUDY DESIGN:
Intervention Model Description: control group and experimental group
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental rehabilitation (Experimental): recived olfactory rehabilitation
  Interventions: Behavioral: olfactory rehabilitation
- control (No Intervention): withouth olfactory rehabilitation

INTERVENTIONS:
Behavioral: olfactory rehabilitation — treatment for improve olfactory function
  Arms: experimental rehabilitation

SUMMARY:
The aim of our study was to compare the recovery of smell in people suffering posttraumatic olfactory impairment following a systematic olfactory rehabilitation performed by occupational therapists to natural recovery in a control posttraumatic group of patients.

DETAILED DESCRIPTION:
Forty participants started the study: 20 for the control group and 20 for the treatment group. The mean of the time span between the traumatic event and the first visit in the rehabilitation group was longer than 22 months, time enough to wait any kind of spontaneous recovery.

In order to establish correct comparisons, the investigators analyzed whether both groups of participants (control group and treatment group) were homogeneous or not regarding the age, gender, time span between the traumatic event and the first visit to the office, brain damage and loss of conscience. Investigators administered visual analogic scale (VAS), CCCRC olfactory test and quality of life questionnaire (RSDI) to both groups at the beginning of the study and 12 months late

ELIGIBILITY:
Inclusion Criteria:

* Olfactory loss participants from institution to the Smell & Tast Office, Otorhinolaryngology Unit, Hospital Universitario Fundación Alcorcón.

All participants provided written informed consent

Exclusion Criteria:

* No sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10-20 (Actual); Primary Completion 2014-10-20 (Actual); Study Completion 2014-10-20 (Actual)

PRIMARY OUTCOMES:
CCCRC | 6 months
  the Connecticut Chemosensorial Clinical Research Centre test (CCCRC) Cain, W.S., Goodspeed, R.B., Gent, J.F. & Leonard, G. (1988). Evaluation of olfactory dysfunction in the Connecticut Clinical Chemosensory Research Centre. Laryngoscope, 98:83-8. https://doi.org/10.1288/00005537-198801000-00017

SECONDARY OUTCOMES:
RSDI | 6 months
  Rhinosinusitis Disability Index. The Rhinosinusitis Disability Index (RSDI) is a 30-item, Likert-scale survey consisting of three individual subscales that include the physical, functional, and emotional domains. Total scores range between 0-120. Higher RSDI total and domain scores imply a higher impact of disease

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No